CLINICAL TRIAL: NCT05690633
Title: Feasibility of Obtaining Pulse Oximetry Readings from the Oropharynx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003039
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Surgery; Arterial Catheterization, Peripheral
MeSH Terms: interventions — Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Oropharyngeal oximetry (Experimental): The use of a pulse oximeter in the oropharynx on either an oral airway or a tongue blade.
  Interventions: Device: Pulse oximetry

INTERVENTIONS:
Device: Pulse oximetry — Noninvasive method of measuring the saturation of oxygen in the blood.

SUMMARY:
This is a prospective study to evaluate the feasibility of obtaining a pulse oximetry ready from the oropharynx with a standard oximeter probe that has been attached to an oral airway or a tongue blade. The study will compare the values from the peripheral pulse oximeter on a finger, toe, foot or hand with the that from the oropharyngeal oximeter. The study will also compare the saturation from an arterial blood gas (ABG) collected as standard of care with that obtained from the oropharyngeal oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a surgical procedure with general anesthesia and requiring an invasive arterial cannula

Exclusion Criteria:

* Patients in whom an arterial cannula is not indicated for the surgical procedure
* Patients in whom a peripheral pulse oximeter value cannot be obtained
* Patients in whom an invasive arterial cannula cannot be placed
* Patients with any type of intra-oral pathology or injury
* Patients in whom access to the oropharynx is restricted or not feasible for any clinical reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Accuracy of Pulse Oximetry | Baseline
  Accuracy of pulse oximetry readings (SpO2) as compared with arterial oxygen saturations

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No